CLINICAL TRIAL: NCT03650569
Title: Italian Angelman Syndrome Registry Protocol
Acronym: RISA
Status: Completed | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1 08.02.2018
Record Dates: First submitted 2018-06-26; First posted 2018-08-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Angelman Syndrome
Keywords: Angelman Syndrome; Caregivers; Parents; Rare diseases; Registries
MeSH Terms: conditions — Angelman Syndrome; Rare Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Italian Angelman Registry is a national registry for patients with Angelman Syndrome. No experimental intervention is involved in participation. The data provided are stored in the registry according the EU General Data Protection Regulation (GDPR, enforced on 25 May 2018), unless participants wish to withdraw their child/ adult's information from the registry.

DETAILED DESCRIPTION:
Parents/caregivers of a child or an adult with Angelman Syndrome living in Italy are eligible to insert data in this registry. The individuals must have a diagnosis of Angelman Syndrome confirmed by genetic testing results. The registry has been launched in February 2018 in coincidence with the International Angelman Day and the recruitment will be open until February 2021.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of Angelman syndrome

Exclusion Criteria:

* Does not meet diagnostic criteria for Angelman Syndrome Other medical or genetic disorders (except autism)

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Angelman syndrome (molecular and clinical diagnosis) from the ages of 1 day onwards
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Medical and behavioral problems | 3 years
  Medical and behavioral problems associated with Angelman syndrome and their prevalence.

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Carriero, Study Director — FROM
Locations (1):
- FROM (Fondazione per la Ricerca Ospedale Maggiore di Bergamo ), Bergamo, Italy

REFERENCES:
- [Background] Augustine EF, Adams HR, Mink JW. Clinical trials in rare disease: challenges and opportunities. J Child Neurol. 2013 Sep;28(9):1142-50. doi: 10.1177/0883073813495959. PMID 24014509
- [Background] Bailus BJ, Segal DJ. The prospect of molecular therapy for Angelman syndrome and other monogenic neurologic disorders. BMC Neurosci. 2014 Jun 19;15:76. doi: 10.1186/1471-2202-15-76. PMID 24946931
- [Background] Bellgard MI, Macgregor A, Janon F, Harvey A, O'Leary P, Hunter A, Dawkins H. A modular approach to disease registry design: successful adoption of an internet-based rare disease registry. Hum Mutat. 2012 Oct;33(10):E2356-66. doi: 10.1002/humu.22154. Epub 2012 Jul 2. PMID 22753342
- [Background] Bi X, Sun J, Ji AX, Baudry M. Potential therapeutic approaches for Angelman syndrome. Expert Opin Ther Targets. 2016;20(5):601-13. doi: 10.1517/14728222.2016.1115837. Epub 2015 Nov 26. PMID 26558806
- [Background] Clayton-Smith J, Laan L. Angelman syndrome: a review of the clinical and genetic aspects. J Med Genet. 2003 Feb;40(2):87-95. doi: 10.1136/jmg.40.2.87. PMID 12566516
- [Background] Gentile JK, Tan WH, Horowitz LT, Bacino CA, Skinner SA, Barbieri-Welge R, Bauer-Carlin A, Beaudet AL, Bichell TJ, Lee HS, Sahoo T, Waisbren SE, Bird LM, Peters SU. A neurodevelopmental survey of Angelman syndrome with genotype-phenotype correlations. J Dev Behav Pediatr. 2010 Sep;31(7):592-601. doi: 10.1097/DBP.0b013e3181ee408e. PMID 20729760
- [Background] Horsler K, Oliver C. The behavioural phenotype of Angelman syndrome. J Intellect Disabil Res. 2006 Jan;50(Pt 1):33-53. doi: 10.1111/j.1365-2788.2005.00730.x. PMID 16316429
- [Background] Laan LA, Halley DJ, den Boer AT, Hennekam RC, Renier WO, Brouwer OF. Angelman syndrome without detectable chromosome 15q11-13 anomaly: clinical study of familial and isolated cases. Am J Med Genet. 1998 Mar 19;76(3):262-8. PMID 9508247
- [Background] Margolis SS, Sell GL, Zbinden MA, Bird LM. Angelman Syndrome. Neurotherapeutics. 2015 Jul;12(3):641-50. doi: 10.1007/s13311-015-0361-y. PMID 26040994
- [Background] Mertz LG, Christensen R, Vogel I, Hertz JM, Ostergaard JR. Eating behavior, prenatal and postnatal growth in Angelman syndrome. Res Dev Disabil. 2014 Nov;35(11):2681-90. doi: 10.1016/j.ridd.2014.07.025. Epub 2014 Jul 26. PMID 25064682
- [Background] Napier KR, Tones M, Simons C, Heussler H, Hunter AA, Cross M, Bellgard MI. A web-based, patient driven registry for Angelman syndrome: the global Angelman syndrome registry. Orphanet J Rare Dis. 2017 Aug 1;12(1):134. doi: 10.1186/s13023-017-0686-1. PMID 28764722
- [Background] Tan WH, Bird LM. Angelman syndrome: Current and emerging therapies in 2016. Am J Med Genet C Semin Med Genet. 2016 Dec;172(4):384-401. doi: 10.1002/ajmg.c.31536. Epub 2016 Nov 8. PMID 27860204
- [Background] Tan WH, Bacino CA, Skinner SA, Anselm I, Barbieri-Welge R, Bauer-Carlin A, Beaudet AL, Bichell TJ, Gentile JK, Glaze DG, Horowitz LT, Kothare SV, Lee HS, Nespeca MP, Peters SU, Sahoo T, Sarco D, Waisbren SE, Bird LM. Angelman syndrome: Mutations influence features in early childhood. Am J Med Genet A. 2011 Jan;155A(1):81-90. doi: 10.1002/ajmg.a.33775. PMID 21204213
- [Background] Tones M, Cross M, Simons C, Napier KR, Hunter A, Bellgard MI, Heussler H. Research protocol: The initiation, design and establishment of the Global Angelman Syndrome Registry. J Intellect Disabil Res. 2018 May;62(5):431-443. doi: 10.1111/jir.12482. PMID 29633452
- [Background] Williams CA, Driscoll DJ, Dagli AI. Clinical and genetic aspects of Angelman syndrome. Genet Med. 2010 Jul;12(7):385-95. doi: 10.1097/GIM.0b013e3181def138. PMID 20445456